CLINICAL TRIAL: NCT04051580
Title: Comparison of Lactated Ringer's Solution and PlasmaLyte-A as a Base Solution for Del Nido Cardioplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 036143
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Myocardial Injury
Keywords: myocardial protection; cardiac surgery; del Nido cardioplegia
MeSH Terms: interventions — Ringer's Lactate; Plasmalyte A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactated Ringer's solution (Experimental): For patients randomized to lactated Ringer's solution (study group), lactated Ringer's solution is used as a base solution for del Nido cardioplegia.
  Interventions: Drug: Lactated Ringer
- PlasmaLyte-A (Active Comparator): For patients randomized to PlasmaLyte-A (control group), PlasmaLyte-A (Baxter Healthcare Corporation, Deerfield, IL, USA) is used as a base solution for del Nido cardioplegia.
  Interventions: Drug: Lactated Ringer

INTERVENTIONS:
Drug: Lactated Ringer — Comparison of Lactated Ringer's Solution and PlasmaLyte-A as a Base Solution for Del Nido Cardioplegia
  Other Names: PlasmaLyte-A

SUMMARY:
Del Nido cardioplegia has been used exclusively for myocardial protection in pediatrics cardiac surgery for decades. Its unique properties including lidocaine which helps counteract potassium depolarization of the myocardial cell membrane, inhibition of intracellular calcium accumulation, preservation of intracellular high-energy phosphates, free-radical scavenging and acid-base buffering have been proven to be very effective for myocardial protection during cardiac surgery for congenital heart disease and acquired heart disease. Recent studies have proven its safety, efficacy, and cost-effectiveness for myocardial protection in adult cardiac surgery as a single dose cardioplegia which is typically administered in a single dose fashion or with extended dosing intervals. In contrast, Traditional blood cardioplegia is commonly administered approximately every 20 minutes. These characteristics of del Nido cardioplegia allow for fewer interruptions and improve surgical workflow. The base solution for del Nido cardioplegia is normally Plasma-Lyte A (Baxter Healthcare Corporation, Deerfield, IL, USA) which has an electrolyte composition similar to the extracellular fluid and is calcium-free. Unfortunately, an unavailability of PlasmaLyte-A in many countries precluding utilization of del Nido cardioplegia with its normal base solution in many cardiac centers. To access the benefits of del Nido cardioplegia, we utilize lactated Ringer's solution as the base solution. This prospective randomized study aimed to evaluate myocardial preservation and clinical outcomes when using lactated Ringer's solution compared with PlasmaLyte-A as a base solution for del Nido cardioplegia.

DETAILED DESCRIPTION:
This clinical trial is performed at Ramathibodi hospital, Mahidol university in Bangkok, Thailand. The protocol has been approved by institutional ethical committee (ref. ID 03-61-43) with informed consent required for all patients.

The difference of 24 hour post-op troponin level between the del Nido cardioplegia and the blood cardioplegia group from previous randomized study were 2.3 (SD 2.1) and 7.0 (SD 14.7) ng/mL, respectively (p = 0.053). Our previous observational study also exhibited comparable results between modified del Nido cardioplegia and blood cardioplegia. The author estimated the sample size of 160 randomized patients to give 80% power at the 5% significant level (alpha 0.05, beta 0.2). Giving allowance for attrition, a sample size of 100 was chosen in each group.

Patients aged 18 years or older undergoing elective cardiac surgery for acquired heart disease (including isolated coronary artery bypass grafting(CABG), isolated valve surgery, combined valve surgery, or concomitant CABG and valve surgery) are randomized 1:1 into lactated Ringer's solution (study group) and PlasmaLyte-A (control group).

For patients randomized to lactated Ringer's solution (study group), lactated Ringer's solution is used as a base solution for del Nido cardioplegia.

For patients randomized to PlasmaLyte-A (control group), PlasmaLyte-A (Baxter Healthcare Corporation, Deerfield, IL, USA) is used as a base solution for del Nido cardioplegia.

Del Nido cardioplegia is delivered 1:4 with 1 part of oxygenated pump blood to 4 parts of cardioplegia solution. Del Nido cardioplegia can be delivered antegrade through aortic root catheter, directly through the coronary ostia or retrograde via the coronary sinus depending on the type of operation and degree of aortic valve insufficiency. Our protocol is to administer a single dose 20 mL/kg with maximum dose of 1000 mL for patients larger than 50 kg. After 90 minutes of aortic cross clamp time, the surgeon decides how much subsequent doses needs to be administered. If coronary bypass grafting is required, 5-10 mL of del Nido cardioplegia is administered via the saphenous vein graft or the radial artery graft to test the distal anastomosis. In our circuit, del Nido cardioplegia passes through a non-recirculating cardioplegia set with a coil heat exchanger and a delivery temperature of 4°C. It is generally administered over 1-2 minutes with system pressure 100-200 mmHg.

Primary outcomes comprised assessments of myocardial injury, including troponin-T level at immediate post-op, 12 hour post-op, and 24 hour post-op.

Secondary outcomes comprised assessments of additional measures of myocardial protection (including incidence of ventricular fibrillation after aortic cross-clamp removal; post-op left ventricular ejection fraction (LVEF) change; duration of inotrope/vasopressor requirement; and requirement for intra-aortic balloon pump (IABP) support), intraoperative outcomes (including total volume of cardioplegia; number of doses; total cardiopulmonary bypass (CPB) time; and aortic cross-clamp time), and clinical outcomes (including intensive care unit ICU) stay; hospital stay; incidence of postoperative atrial fibrillation or flutter; mortality; postoperative complications; and red cell transfusion).

Patient characteristics and postoperative outcomes were as defined by the Society of Thoracic Surgeons (STS) Adult Cardiac Surgical Database. LVEF was assessed by transesophageal echocardiography before surgery and at the end of operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years or older undergoing elective adult cardiac surgery

Exclusion Criteria:

* Emergency surgery
* Patient who does not want to participate in the study
* Lidocaine allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Myocardial injury | 24 hour post-op
  troponin-T level at 24 hour post-op

SECONDARY OUTCOMES:
Incidence of ventricular fibrillation after aortic cross-clamp removal | Intra-operative period
  Ventricular fibrillation after aortic cross-clamp removal required defibrillation
Post-op left ventricular ejection fraction (LVEF) change | Intra-operative period
  Difference between pre-op and post-op LVEF. LVEF was assessed by transesophageal echocardiography before surgery and at the end of operation.
Duration of inotrope/vasopressor requirement | up to 1 hour (During admission in intensive care unit)
  Length of inotropic or vasopressor support in intensive care unit (hour)
Incidence of intra-aortic balloon pump (IABP) insertion | up to 1 hour (During admission in intensive care unit)
  Requirement for intra-aortic balloon pump (IABP) support
Incidence of Operative mortality | up to 1 month postoperatively
  Operative mortality includes both (1) all deaths occurring during the hospitalization in which the operation was performed, even if after 30 days; and (2) those deaths occurring after discharge from the hospital, but within 30 days of the procedure.
Incidence of Permanent Stroke | up to 1 month postoperatively
  Postoperative stroke (i.e., any confirmed neurological deficit of abrupt onset caused by a disturbance in blood supply to the brain that did not resolve within 24 hours.
Incidence of Renal Failure | up to 1 month postoperatively
  Acute or worsening renal failure resulting in one or more of the following:1.Increase of serum creatinine to ≥ 4.0 with an increase of at least 0.5mg/dl or 3x most recent preoperative creatinine level.2.A new requirement for dialysis postoperatively.
Incidence of Prolonged Ventilation > 24 hours | up to 1 month postoperatively
  Prolonged post-operative pulmonary ventilation > 24.0 hours. The hours of postoperative ventilation time include OR exit until extubation, plus any additional hours following reintubation.
Incidence of Deep sternal wound infection | up to 1 month postoperatively
  Deep sternal wound infection or mediastinitis (according to CDC definition) diagnosed within 30 days of the operation or any time during the hospitalization for the surgery
Incidence of Reoperation for any reason | up to 1 month postoperatively
  Reoperation for bleeding/tamponade, valvular dysfunction, graft occlusion, other cardiac reason, or non-cardiac reason
Incidence of Major Morbidity or Operative Mortality | up to 1 month postoperatively
  A composite endpoint defined as any of the outcomes listed above, including; Operative mortality, Permanent Stroke,Renal Failure, Prolonged Ventilation > 24 hours, Deep sternal wound infection, Reoperation for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Narongrit Kantathut, MD, Principal Investigator — Ramathibodi hospital, Mahidol University
Locations (1):
- Ramathibodi Hospital, Bangkok, Thailand

REFERENCES:
- [Background] Ad N, Holmes SD, Massimiano PS, Rongione AJ, Fornaresio LM, Fitzgerald D. The use of del Nido cardioplegia in adult cardiac surgery: A prospective randomized trial. J Thorac Cardiovasc Surg. 2018 Mar;155(3):1011-1018. doi: 10.1016/j.jtcvs.2017.09.146. Epub 2017 Nov 13. PMID 29246552
- [Result] Kantathut N, Krathong P, Khajarern S, Leelayana P, Cherntanomwong P. Comparison of lactated Ringer's solution and Plasma-Lyte A as a base solution for del Nido cardioplegia: a prospective randomized trial. Eur J Cardiothorac Surg. 2024 Mar 1;65(3):ezae018. doi: 10.1093/ejcts/ezae018. PMID 38244592